CLINICAL TRIAL: NCT01144741
Title: Study of Therapeutic Outcomes and Practices in Freeman-Sheldon Syndrome
Brief Title: Survey Study and Records Review of Treatment Outcomes in Freeman-Sheldon Syndrome
Acronym: STOP-FSS
Status: Terminated | Type: Observational
Why Stopped: Insufficient patient enrolment
Sponsor: Freeman-Sheldon Research Group, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 000063; U1111-1120-5851 (Other: World Health Organisation, Universal Trial Number)
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Freeman-Sheldon Syndrome; Arthrogryposis Distal Type 2A; Whistling Face Syndrome; Craniocarpotarsal Dysplasia; Craniocarpotarsal Dystrophy; Freeman-Sheldon Syndrome Variant; Sheldon-Hall Syndrome; Arthrogryposis Distal Type 2B; Gordon Syndrome; Arthrogryposis Distal Type 3; Arthrogryposis Distal Type 1; Arthrogryposis, Distal, Type 1A; Arthrogryposis Distal Type 1B; Arthrogryposis, Distal; Craniofacial Abnormalities; Arthrogryposis
Keywords: rehabilitation; surgery; therapy; Quality Of Life; Health-Related Quality Of Life; Health Status; Depressive Symptoms; Situational Depression
MeSH Terms: conditions — Freeman-Sheldon syndrome; Distal arthrogryposis type 2B; Gordon syndrome; Pseudohypoaldosteronism; Digitotalar Dysmorphism; Arthrogryposis; Craniofacial Abnormalities; Depression | interventions — Multicenter Studies as Topic; Metabolism; Health Records, Personal; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Any specimens received as part of records review, such as pathology microscope slides or frozen sections, will be retained as per institutional policy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Freeman-Sheldon syndrome Classic Type: Patients who have all features required by the Stevenson criteria, including: very small mouth (microstomia); whistling-face appearance (pursed lips); "H" or "V" shaped chin dimple; very obvious down-slanting crease from the nostril to the corners of the mouth (nasolabial creases); and restricted movement in joints (contractures) of two or more body areas, often hands and feet, with fingers and toes frequently overlapping.
  Interventions: Other: PTSD Checklist-Civilian (PCL-C); Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale (CES-D); Other: Functional Enquiry (or Review of Systems) Form; Other: Study of Therapeutic Outcomes and Practices in Freeman-Sheldon Syndrome (STOP-FSS) Questionnaire; Other: FSRG Semi-Structured Quality of Life Interview (FSRG SSQLI); Other: Medical Records Review
- Freeman-Sheldon syndrome Craniofacial Type: Patients who have only the face and skull physical findings required by the Stevenson criteria, including: very small mouth (microstomia), whistling-face appearance (pursed lips), "H" or "V" shaped chin dimple, very obvious down-slanting crease from the nostril to the corners of the mouth (nasolabial creases).
  Interventions: Other: PTSD Checklist-Civilian (PCL-C); Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale (CES-D); Other: Functional Enquiry (or Review of Systems) Form; Other: Study of Therapeutic Outcomes and Practices in Freeman-Sheldon Syndrome (STOP-FSS) Questionnaire; Other: FSRG Semi-Structured Quality of Life Interview (FSRG SSQLI); Other: Medical Records Review
- Freeman-Sheldon syndrome Mixed Type: Patients who have the face and skull physical findings required by the Stevenson criteria and some but not all required joint problems.
  Interventions: Other: PTSD Checklist-Civilian (PCL-C); Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale (CES-D); Other: Functional Enquiry (or Review of Systems) Form; Other: Study of Therapeutic Outcomes and Practices in Freeman-Sheldon Syndrome (STOP-FSS) Questionnaire; Other: FSRG Semi-Structured Quality of Life Interview (FSRG SSQLI); Other: Medical Records Review
- Sheldon-Hall syndrome: Patients who have all features required by the Stevenson criteria, including: small mouth (not microstomia); neck webbing (pterygium colli); small but prominent chin; very obvious down-slanting crease from the nostril to the corners of the mouth (nasolabial creases); and restricted movement in joints (contractures) of two or more body areas, often hands and feet, with fingers and toes frequently overlapping.
  Interventions: Other: PTSD Checklist-Civilian (PCL-C); Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale (CES-D); Other: Functional Enquiry (or Review of Systems) Form; Other: Study of Therapeutic Outcomes and Practices in Freeman-Sheldon Syndrome (STOP-FSS) Questionnaire; Other: FSRG Semi-Structured Quality of Life Interview (FSRG SSQLI); Other: Medical Records Review
- Distal Arthrogryposis Type 1: Patients with features consistent with this diagnosis, including restricted movement in joints (contractures) of two or more body areas, often hands and feet, with fingers and toes frequently overlapping.
  Interventions: Other: PTSD Checklist-Civilian (PCL-C); Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale (CES-D); Other: Functional Enquiry (or Review of Systems) Form; Other: Study of Therapeutic Outcomes and Practices in Freeman-Sheldon Syndrome (STOP-FSS) Questionnaire; Other: FSRG Semi-Structured Quality of Life Interview (FSRG SSQLI); Other: Medical Records Review
- Distal Arthrogryposis Type 3: Patients with features consistent with this diagnosis, including: gap in the roof of the mouth (cleft palate); drooping eyelid (blepharoptosis); and backbones curve problems; and restricted movement in joints (contractures) of two or more body areas, often hands and feet, with fingers and toes frequently overlapping.
  Interventions: Other: PTSD Checklist-Civilian (PCL-C); Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale (CES-D); Other: Functional Enquiry (or Review of Systems) Form; Other: Study of Therapeutic Outcomes and Practices in Freeman-Sheldon Syndrome (STOP-FSS) Questionnaire; Other: FSRG Semi-Structured Quality of Life Interview (FSRG SSQLI); Other: Medical Records Review

INTERVENTIONS:
Other: PTSD Checklist-Civilian (PCL-C) — Completed by patients before the interview; it is a 17-item survey listing of symptoms of posttraumatic stress disorder.
Other: Modified Flanagan Quality of Life Scale — Completed by patients before the interview; it is a 16-item survey designed for use in persons with chronic illness.
  Other Names: Quality of Life Scale; Quality of Life Instrument; Quality of Life Measure
Other: Center for Epidemiologic Studies Depression Scale (CES-D) — Completed by patients before the interview; it is a 20-item survey that asks about depressive feelings and behaviours in the past week.
Other: Functional Enquiry (or Review of Systems) Form — Completed during the interview; it is a checklist of medical problems.
  Other Names: Health History; Systems Review; Medical History
Other: Study of Therapeutic Outcomes and Practices in Freeman-Sheldon Syndrome (STOP-FSS) Questionnaire — The STOP Questionnaire is a guided interview form that will be used to assess diagnosis, problems, treatments, and outcomes.
Other: FSRG Semi-Structured Quality of Life Interview (FSRG SSQLI) — Completed after data analysis from the existing surveys, it will be a specific quality of life interview, taking into consideration individual's total health outcome.
  Other Names: Quality of Life Assessment; quality of life instrument; quality of life measure
Other: Medical Records Review — Review of medical records will be used, along with STOP-FSS Survey to assess patient histories and outcomes.
  Other Names: Treatment Records Review; Review of Patient Notes; Patient Chart Review; Review of Clinical Data

SUMMARY:
Freeman-Sheldon syndrome (FSS) is a rare muscle disorder present before birth, involving primarily problems of the face and skull and the hands and feet.

This is a study of problems, experiences, helpful treatments, and quality of life focusing on patients with FSS but including patients with Sheldon-Hall syndrome (SHS), distal arthrogryposis type 1 (DA1), and distal arthrogryposis type 3 (DA3), also called Gorden syndrome. These and related disorders are very challenging to treat, partly because the big differences in individual patients and lack of information on previous clinical experience with treatment options. It is hoped the study will identify areas for further research in physiology and therapy.

This study will cover all types of treatment [medical (non-surgical), including psychiatric, and surgical treatments], even unconventional. It also includes questions about effects on the patient's thoughts, feelings, quality of life, and relationship with siblings, family, and parents' and if any intervention was required or advised. This study will also look for similarities and differences in patients who meet the head and face part of the diagnostic criteria but do not meet all other parts and patients who met the full diagnostic criteria. There will be questions about problems or experiences to investigate if both groups of patients may have the same syndrome. Treatment success depends on getting a correct diagnosis.

DETAILED DESCRIPTION:
This study was initiated by the research assistant (Mikaela I. Poling) and assisted by another research assistant (J. Andrés Morales), as part of their academic project on these syndromes, under the supervision of the Principal Investigator (Robert L Chamberlain).

Classic FSS, SHS, DA1, and DA3 are poorly understood pathological entities that share some similar physical findings to FSS. Stevenson et al. (2006) provided the only study to date on FSS features and history. They did not, however, focus on therapeutic outcomes, and there was limited anecdotal outcome data in single and multiple case reports.

The objectives for STOP-FSS are as follows: to evaluate (1) physical findings, possible frequency clusters, and complications of physical findings amongst patients with FSS; (2) posttraumatic stress and depressive symptoms and associated therapeutic outcomes in patients with FSS, using single-disease specific (i.e., posttraumatic stress symptoms, chronic depression) measures; (3) document treatment types and outcomes; (4) evaluate quality of life in patients with FSS, using a general quality of life self-report measure and syndrome-specific semi-structured quality of life interview; (5) educational attainment and services used; (6) evaluate diagnostic accuracy of FSS and SHS, using the Stevenson criteria; and (7) evaluate possible differences with patients meeting the full Stevenson criteria and those fulfilling the craniofacial part of the Stevenson criteria, with or without additional malformations.

The following hypotheses are thus proposed. First, it is suggested that physical findings and frequency clusters will be similar to those previously reported, but complications of physical findings amongst patients with FSS, having received little attention in the literature, will be pronounced and result in nearly as significant of a disease burden for the patient as the primary physical findings themselves, e.g., intercostal myopathy eventually leading to right heart failure in some patients. Second, it is suggested that FSS is associated with higher rates of posttraumatic stress symptoms, depressive symptoms than is observed in the general population. Third, it is suggested that physiotherapy alone or with surgery is expected to be superior to surgery alone, especially for patients with FSS, in treating most problems, but surgery may have an important role, especially treating blepharophimosis and in combination with intensive pre- and post-operative physiotherapy in treating selective tendon lengthening in hands and feet. Fourth, it is suggested that FSS is associated with reduced quality of life than is observed in the general population. Fifth, it is suggested that when patients with FSS who do not have neurocognitive features receive the appropriate academic services, they frequently excel beyond family and peers, and it is also suggested that most patients with FSS do not receive educational services that are responsive to their unique needs and abilities, e.g., placement in 'special' classes or schools based on the patient's appearance or poorly conducted intelligence tests. Sixth, it is suggested, based on systematic review and meta-analysis preliminary results, that two-thirds of patients with a stated diagnosis of FSS will not meet the Stevenson criteria and be rediagnosed, mostly as DA1. Seventh, it is suggested, based on systematic review and meta-analysis preliminary results, that two-thirds of patients with stated diagnosis of FSS who do not meet the Stevenson criteria, one-third will be meet the craniofacial stipulates of the Stevenson criteria, with or without additional malformations, and share a natural history with those who met the full Stevenson criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have phenotypes consistent with (1) the Stevenson criteria for classic FBS or SHS; (2) one of four tentative FBS subtypes; or (3) DA1A, DA1B, or DA3.
* Any of the following: (1) patients or parents of minor children willing to give consent, or (2) patients who are deceased or (3) retrospective chart review patients (living or deceased) who have enough clinical data available to establish the diagnosis and satisfy minimum data collection requirements.
* Persons who speak English, Spanish, German, Russian, or Czech.

Exclusion Criteria:

* Patients who do not have phenotypes consistent with (1) the Stevenson criteria for classic FBS or SHS; (2) one of four tentative FBS subtypes; or (3) DA1A, DA1B, or DA3.
* Any of the following: (1) patients or parents of minor children not willing to give consent, or (2) patients who are deceased or (3) retrospective chart review patients (living or deceased) who do not have enough clinical data available to establish the diagnosis and satisfy minimum data collection requirements.
* Potentially persons who speak languages other than English, Spanish, German, Russian, or Czech, subject to translator availability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There are no patient enrollment restrictions based on gender, ethnicity, religion, socio-economic status, geographical location, or clinical setting.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Physical Findings and Complications of Physical Findings | during a single study interview, which lasts 1-2 hours
  The frequency to which certain features of the syndromes contribute to mortality or morbidity, especially life-long functional impairment.

SECONDARY OUTCOMES:
Posttraumatic Stress and Depressive Symptoms | at study enrolment and during a single study interview, which lasts 1-2 hours
  Increased frequency of mental health symptoms (posttraumatic and depressive) over expected for general population

OTHER OUTCOMES:
Intervention-Related Outcome | during a single study interview, which lasts 1-2 hours
  Self-report or medical record evidence of ability to complete activities of daily living and instrumental activities of daily living compared with abilities before each intervention reported and, if relevant, how long this change in abilities lasted
Quality of Life Status | at enrolment and during a single study interview, which lasts 1-2 hours
  Stated and evidenced experience of life
Educational attainment | during a single study interview, which lasts 1-2 hours
  Educational level completed compared with age
Diagnostic Accuracy for Freeman-Sheldon and Sheldon-Hall syndromes | at study enrolment
  Correct diagnosis, using the Stevenson criteria
Correlations of Full and Partial Stevenson Criteria Freeman-Sheldon syndrome with | at study enrolment and during a single study interview, which lasts 1-2 hours
  Significant differences or correlations of patients meeting the full Stevenson criteria for FSS with those fulfilling the craniofacial part of the Stevenson criteria, with or without additional malformations

CONTACTS AND LOCATIONS:
Locations (1):
- Freeman-Sheldon Research Group, Inc. Headquarters, Buckhannon, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared, due to concerns involved in masking identities of individuals with such a rare condition.

REFERENCES:
- [Background] Poling MI, Morales Corado JA, Chamberlain RL. Findings, phenotypes, and outcomes in Freeman-Sheldon and Sheldon-Hall syndromes and distal arthrogryposis types 1 and 3: protocol for systematic review and patient-level data meta-analysis. Syst Rev. 2017 Mar 6;6(1):46. doi: 10.1186/s13643-017-0444-4. PMID 28264711
- [Result] Chamberlain RL, Poling MI, Portillo AL, Morales A, Ramirez RR, McCormick RJ. Freeman-Sheldon syndrome in a 29-year-old woman presenting with rare and previously undescribed features. BMJ Case Rep. 2015 Oct 22;2015:bcr2015212607. doi: 10.1136/bcr-2015-212607. PMID 26494722